CLINICAL TRIAL: NCT06347822
Title: Implementation of Single Session Interventions in Integrated Behavioral Health: Increasing Access to Evidence-based Care
Brief Title: Increasing Access to Evidence-Based Care in Integrated Behavioral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anne I. Roche, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-011276
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Session Therapy Visit (Experimental): Subjects will have a single-session therapy visit with an Integrated Behavioral Health (IBH) clinician.
  Interventions: Behavioral: Therapy Session

INTERVENTIONS:
Behavioral: Therapy Session — Single-session intervention (SSI) based on acceptance and commitment therapy (ACT) and solution-focused brief therapy (SFBT) principles

SUMMARY:
The purpose of this research is to explore whether a single-session therapy visit may be of interest to patients seeking mental health services in Mayo Clinic's Integrated Behavioral Health program and whether a single-session therapy visit may be helpful in improving mental health. Researchers hope to better understand whether single-session visits could be a helpful option to offer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient currently scheduled for an IBH consultation session at Mayo Clinic Rochester.
* Able to read and speak English.

Exclusion Criteria:

* Individuals diagnosed with psychotic spectrum, Bipolar I and II, or severe substance use disorder and individuals with severe cognitive impairment per chart review will not be eligible and will not be contacted about the study. Individuals must score ≥ 5 on the PHQ-9 and/or GAD-7 but not >14 on either measure (indicating mild to moderate depression and/or anxiety) and respond < 2 to Item 9 of the PHQ-9 ("thoughts that you would be better off dead, or thoughts of hurting yourself in some way") to be eligible for the study.
* Patients who are ineligible will remain scheduled for a regular IBH therapy consultation as originally planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction with IBH therapy | Immediately post-intervention (1-1.25 hours after study visit initiation)
  Measured using the Client Satisfaction Questionnaire-8 (CSQ-8). Total scores range from 8 to 32, with higher number indicating greater satisfaction.
Satisfaction with Action Plan | Immediately post-intervention (1-1.25 hours after study visit initiation)
  We will use 3 items rated on a five-point scale (0 = not at all, 4 = very much) to assess participant satisfaction with their Action Plan ("Did the visit help you develop an action plan?"; "How hopeful are you that the action plan will be useful?" and "How motivated do you feel to use your action plan?"). Scores will range from 0-12 with higher scores indicating greater satisfaction with the Action Plan.
Change in readiness for change scores | Baseline and immediately post-intervention (1-1.25 hours after study visit initiation)
  The readiness for change ruler is a 3 item measure that examines participant's willingness to change to improve their mental health on a 0 (not at all confident/important/ready) to 10 scale (completely confident/important/ready). The total score ranges from 0 to 30, with higher scores indicating higher levels of willingness to change.
Change in belief in capacity to generate routes to reach goals (pathways) | Baseline and immediately post-intervention (1-1.25 hours after study visit initiation)
  The State Hope Scale (Pathways subscale) is a 3 item measure that assesses participant belief in their capacity to generate routes to reach goals. Scale responses range from 1 (Definitely false) to 8 (Definitely true), with total scores ranging from 3-24 and higher scores indicating higher levels of pathways thinking.
Change in PHQ-9 scores | Baseline and 2-week follow-up
  The PHQ-9 asks participants to rate 9 questions assessing dimensions of depression on a scale of 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 27 with higher scores indicating higher levels of depression.
Change in GAD-7 scores | Baseline and 2-week follow-up
  The GAD-7 asks participants to rate 7 statements based on how generally anxious they have felt over the past 2 weeks on a 4 point scale ranging from 0 (Not at all) to 3 (Nearly every day). Total score ranges from 0 to 21 with higher scores representing higher generalized anxiety.

SECONDARY OUTCOMES:
Change in Valuing Questionnaire (Values Progress subscale) | Baseline and 2-week follow-up
  The 10-item Valuing Questionnaire asks participants to rate statements about valued living on a 7-point Likert-type scale ranging from 0 (not at all true) to 6 (completely true). The measure assesses two subscales, Values Progress (0-30) and Values Obstruction (0-30), with higher scores on each indicating greater values progress and obstruction, respectively.
Change in Valuing Questionnaire (Values Obstruction subscale) | Baseline and 2-week follow-up
  The 10-item Valuing Questionnaire asks participants to rate statements about valued living on a 7-point Likert-type scale ranging from 0 (not at all true) to 6 (completely true). The measure assesses two subscales, Values Progress (0-30) and Values Obstruction (0-30), with higher scores on each indicating greater values progress and obstruction, respectively.
Change in CompACT scores (Valued Action) | Baseline and 2-week follow-up
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes-15 item (CompACT) is used to assess psychological flexibility (three subscales of openness to experience, behavioral awareness, and valued action). Each item is rated on a scale of 0 to 6 (0 = strongly disagree, 6 = strongly agree). Higher scores on each subscale (VA, OE, BA) indicate greater valued action (VA), greater openness to experience (OE), and greater behavioral awareness (BA), respectively.
Change in CompACT scores (Openness to Experience) | Baseline and 2-week follow-up
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes-15 item (CompACT) is used to assess psychological flexibility (three subscales of openness to experience, behavioral awareness, and valued action). Each item is rated on a scale of 0 to 6 (0 = strongly disagree, 6 = strongly agree). Higher scores on each subscale (VA, OE, BA) indicate greater valued action (VA), greater openness to experience (OE), and greater behavioral awareness (BA), respectively.
Change in CompACT scores (Behavioral Awareness) | Baseline and 2-week follow-up
  The Comprehensive Assessment of Acceptance and Commitment Therapy Processes-15 item (CompACT) is used to assess psychological flexibility (three subscales of openness to experience, behavioral awareness, and valued action). Each item is rated on a scale of 0 to 6 (0 = strongly disagree, 6 = strongly agree). Higher scores on each subscale (VA, OE, BA) indicate greater valued action (VA), greater openness to experience (OE), and greater behavioral awareness (BA), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Roche, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No